CLINICAL TRIAL: NCT02022748
Title: A Single Dose, Randomized, Open-Label, Parallel Group Study Comparing the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Ticagrelor in Hemodialysis Patients to Subjects With Normal Renal Function
Brief Title: Pharmacokinetics, Pharmacodynamics, and Safety Study of Ticagrelor in Hemodialysis Patients and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5130L00067
Record Dates: First submitted 2013-12-22; First posted 2013-12-30 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): hemodialysis patients: subjects will receive treatment A (ticagrelor oral 90 mg 1 day following the dialysis session but 2 days before the next dialysis session) in period 1 and treatment B (ticagrelor oral 90 mg just prior to dialysis session) in period 2.
  Interventions: Drug: ticagrelor
- Sequence 2 (Experimental): hemodialysis patients: subjects will receive treatment B (ticagrelor oral 90 mg just prior to dialysis session) in period 1 and treatment A (ticagrelor oral 90 mg 1 day following the dialysis session but 2 days before the next dialysis session) in period 2.
  Interventions: Drug: ticagrelor
- Treatment H (Experimental): Healthy subjects: ticagrelor oral 90 mg on 1 day of treatment
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: ticagrelor — Group A is hemodialysis subjects. Crossover design will be implemented for Group A subjects. Group A will be randomized into 2 sequences, Sequence 1 and Sequence 2. In Sequence 1, subjects will receive treatment A in Period 1 and treatment B in Period 2. Washout period of at least 7 days between Period 1 and Period 2 in Sequence 1. Treatment A and Treatment B are defined as follows: Treatment A subjects will be dosed with oral 90 mg ticagrelor tablet 1 day following the dialysis session but 2 days before the next dialysis session. Treatment B will be dosed with oral 90 mg ticagrelor tablet just prior to dialysis session.
  Other Names: Brilinta
  Arms: Sequence 1
Drug: ticagrelor — Group A is hemodialysis subjects. Crossover design will be implemented for Group A subjects. Group A will be randomized into 2 sequences, Sequence 1 and Sequence 2. In Sequence 2, subjects will receive treatment B in Period 1 and treatment A in Period 2. Washout period of at least 7 days between Period 1 and Period 2 in Sequence 2. Treatment A and Treatment B are defined as follows: Treatment A subjects will be dosed with oral 90 mg ticagrelor tablet 1 day following the dialysis session but 2 days before the next dialysis session. Treatment B will be dosed with oral 90 mg ticagrelor tablet just prior to dialysis session.
  Other Names: Brilinta
  Arms: Sequence 2
Drug: ticagrelor — Group B is healthy subjects. Group B healthy subjects will receive oral 90 mg ticagrelor referred to as Treatment H.
  Other Names: Brilinta
  Arms: Treatment H

SUMMARY:
A phase I, open-label study comparing the pharmacokinetics, pharmacodynamics, safety and tolerability of ticagrelor in hemodialysis patients to healthy subjects with normal renal function.

DETAILED DESCRIPTION:
This will be a single dose, randomised, open label, parallel group study conducted in the US to examine the Pharmacokinetics (PK), Pharmacodynamics (PD), safety, and tolerability of ticagrelor in end stage renal disease (ESRD) subjects on hemodialysis (HD) compared with healthy subjects with normal renal function. Up to a total of 30 male and female adult subjects aged 18 to 80 years (inclusive) with a weight of at least 50 kg and a body mass index between 18 and 40 kg/m2 (inclusive), will be dosed to assure that there will be 20 evaluable subjects (10 subjects on HD and in 10 healthy subjects with normal renal function (CrCL ≥90 mL/min). The normal renal function groups should have a similar distribution with respect to age, weight and gender. Subjects will be required to have an inpatient stay from the day prior to dosing until the 48-hour post-dose time-point to ensure that all PK samples are collected at the appropriate timepoints. The study will be conducted in two groups: Group A consisting of ESRD subjects on HD, Group B consisting of healthy subjects. A crossover design will be implemented for Group A subjects as follows: Group A subjects will be randomized into two sequences, Sequence 1 and Sequence 2. In Sequence 1, subjects will receive treatment A in Period 1 and treatment B in Period 2. There will be washout period of at least 7 days between Period 1 and Period 2 in Sequence 1. Similarly in Sequence 2, subjects will receive treatment B in Period 1 and treatment A in Period 2. There will be a washout period of at least 7 days between Period 1 and Period 2 in Sequence 2 as well. Treatment A and treatment B are defined as follows: Treatment A: subjects will be dosed with an oral 90 mg ticagrelor tablet 1 day following the dialysis session but 2 days before the next dialysis session; • Treatment B: subjects will be dosed with an oral 90 mg ticagrelor tablet just prior to dialysis session.(NB: Treatment B dosing should occur within 5 minutes of dialysis start). Group B subjects (healthy subjects) with normal renal function (CrCL of ≥ 90 mL/min) will receive just an oral 90 mg ticagrelor referred to as treatment H. All doses will be administered in an open-label design.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18 to 80 years (inclusive).
* Normal renal function (CrCl of ≥90 mL/min) or End Stage Renal Disease (ESRD) requiring hemodialysis.

Exclusion Criteria:

* Any indication for oral anticoagulant or anti platelet treatment during study period. Must be off treatment for at least 3 weeks (low dose 81mg aspirin is allowed for hemodialysis subjects only).
* Acute Coronary Syndrome (ACS) within past 12 months.
* Contraindications to ticagrelor (ie: active pathological bleeding, severe hepatic impairment, history of hemorrhagic stroke, allergic to ticagrelor).
* Platelet count <100000/μL, hemoglobin <9g/dL
* Blood donation within 90 days of dosing
* Risk for bradycardia
* Investigational drug within 30 days or 6 half-lives, whichever is longer, before dosing
* Concomitant therapy with CYP3A inhibitors/substrates with narrow therapeutic index,or strong CYP3A inducers 14 days before dosing until completion of the follow-up visit.
* History of alcohol, drug, or substance abuse within the past year
* Clinically significant laboratory abnormalities as judged by the investigator.
* Increased bleeding risk including GI bleeding in past 30 days; history of intracranial, retroperitoneal, or spinal bleeding, recent major trauma within 30 days of dosing, Sustained uncontrolled hypertension, history of hemorrhagic disorders.
* Pregnant or lactating females, or females of child-bearing potential (ie, those who are not chemically or surgically sterilised or who are not post-menopause) who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator throughout the duration of the study OR females who have a positive pregnancy test at Visit 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-12-29 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2016-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolene K Berg, MD, Principal Investigator — DaVita Clinical Research, Minneapolis, MN
Locations (2):
- United States (2):
  - Research Site, Lakewood, Colorado
  - Research Site, Minneapolis, Minnesota

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 56 subjects signed ICF, 34 Hemodialysis (HD) subjects and 22 Healthy subjects (HS) at 2 study centers in the US. 27 subjects received treatment (14 HD and 13 HS). First patient signed ICF on 29 December 2013. Due to protocol amendment, the first patient was randomized 22 months later on 20 October 2015, last patient last visit was 09 May 2016.
Pre-assignment Details: 21 out of 34 HD subjects were randomized (13 failed to fulfill eligibility criteria) and 14 were eligible after eligibility re-assessment (5 no longer met the eligibility criteria and 2 experienced Adverse Events (AE) prior to treatment). 13 out of 22 HS were eligible to be treated (9 failed to meet the eligibility criteria).
Groups:
- Sequence 1 (AB): hemodialysis patients: subjects will receive treatment A (ticagrelor oral 90 mg 1 day following the dialysis session but 2 days before the next dialysis session) in period 1 and treatment B (ticagrelor oral 90 mg just prior to dialysis session) in period 2.
- Sequence 2 (BA): Hemodialysis patients: subjects will receive treatment B (ticagrelor oral 90 mg just prior to dialysis session) in period 1 and treatment A (ticagrelor oral 90 mg 1 day following the dialysis session but 2 days before the next dialysis session) in period 2.
Period: Overall Study
Arm/Group | Sequence 1 (AB) | Sequence 2 (BA) | Treatment H
Started | 8 | 6 | 13
Subject Who Started Treatment | 8 | 6 | 13
Subjects Who Completed Treatment | 7 | 4 | 13
Completed | 7 | 4 | 13
Not Completed | 1 | 2 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All 14 randomized HD subjects after eligibility re-assessment (8 in Sequence 1 (AB) and 6 in Sequence 2 (BA)) and 13 eligibile HS are used for baseline analysis.
Groups:
- HD Subjects: Hemodialysis subjects
- HS Subjects: Healthy subjects
- Total: Total of all reporting groups
Arm/Group | HD Subjects | HS Subjects | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (12.5) | 43.8 (10.4) | 47.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 12 | 10 | 22
Weight [Mean (Standard Deviation); unit: kg] | 85.1 (18.3) | 89.0 (16.2) | 87.0 (17.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.77 (4.18) | 28.27 (3.75) | 28.01 (3.91)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter Cmax of Ticagrelor
Time Frame: 0, 1, 2, 4, 6, 12, 24, 36, 48 hours post-dose
Population: The Pharmacokinetic (PK) analysis set included all subjects who received at least 1 dose of study medication and for whom PK data are available with no major protocol deviations thought to significantly affect the pharmacokinetics of ticagrelor or its active metabolite AR-C124910XX.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment A: HD subjects were dosed with an oral 90 mg ticagrelor tablet 1 day following the dialysis session but 2 days before the next dialysis session;
- Treatment B: HD subjects were dosed with an oral 90 mg ticagrelor tablet just prior to dialysis session.
- Treatment H: Healthy subjects (HS) with normal renal function (CrCL of ≥90 mL/min) received one oral 90 mg ticagrelor tablet
Arm/Group | Treatment A | Treatment B | Treatment H
Number analyzed (Participants) | 12 | 13 | 13
ng/mL | 560.32 (54.0) | 598.35 (47.9) | 370.76 (37.3)
Statistical Analysis 1: Comparison: Treatment A vs Treatment H; Test type: Other; Ratio of Geometric Least Square Means = 151.13, 90% CI 2-sided [112.03 to 203.86] — Treatment H is the reference treatment
Statistical Analysis 2: Comparison: Treatment B vs Treatment H; Test type: Other; Ratio of Geometric Least Square Means = 161.38, 90% CI 2-sided [122.52 to 212.58] — Treatment H is the reference treatment
Statistical Analysis 3: Comparison: Treatment A vs Treatment B; Test type: Other; Ratio of Geometric Least Square Means = 90.10, 90% CI 2-sided [78.07 to 103.98] — A linear mixed model with sequence, period, and treatment as fixed effects, and subject-within-sequence as a random effect, was used to analyze the natural log-transformed values of the PK parameters. Treatment B is the reference treatment

2. Primary Outcome: Pharmacokinetic Parameter Cmax of AR-C124910XX
Time Frame: 0, 1, 2, 4, 6, 12, 24, 36, 48 hours post-dose
Population: The PK analysis set included all subjects who received at least 1 dose of study medication and for whom PK data are available with no major protocol deviations thought to significantly affect the pharmacokinetics of ticagrelor or its active metabolite AR-C124910XX.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment H
Number analyzed (Participants) | 12 | 13 | 13
ng/mL | 130.82 (38.3) | 152.25 (54.3) | 111.73 (60.0)
Statistical Analysis 1: Comparison: Treatment A vs Treatment H; Test type: Other; Ratio of Geometric Least Square Means = 117.09, 90% CI 2-sided [84.51 to 162.22] — Treatment H is the reference treatment
Statistical Analysis 2: Comparison: Treatment B vs Treatment H; Test type: Other; Ratio of Geometric Least Square Means = 136.27, 90% CI 2-sided [95.38 to 194.70] — Treatment H is the reference treatment
Statistical Analysis 3: Comparison: Treatment A vs Treatment B; Test type: Other; Ratio of Geometric Least Square Means = 82.29, 90% CI 2-sided [68.43 to 98.96] — [estimate comment as in outcome 1, analysis 3]

3. Primary Outcome: Pharmacokinetic Parameter AUC0-∞ (Area Under the Plasma Concentration-time Curve From Time Zero to Infinity) of Ticagrelor
Time Frame: 0, 1, 2, 4, 6, 12, 24, 36, 48 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A | Treatment B | Treatment H
Number analyzed (Participants) | 12 | 13 | 13
ng*h/mL | 3015.1 (54.2) | 3256.1 (52.5) | 2188.8 (22.6)
Statistical Analysis 1: Comparison: Treatment A vs Treatment H; Test type: Other; Ratio of Geometric Least Square Means = 137.75, 90% CI 2-sided [105.70 to 179.52] — Treatment H is the reference treatment
Statistical Analysis 2: Comparison: Treatment B vs Treatment H; Test type: Other; Ratio of Geometric Least Square Means = 148.76, 90% CI 2-sided [115.07 to 192.32] — Treatment H is the reference treatment
Statistical Analysis 3: Comparison: Treatment A vs Treatment B; Test type: Other; Ratio of Geometric Least Square Means = 90.35, 90% CI 2-sided [77.55 to 105.27] — [estimate comment as in outcome 1, analysis 3]

4. Primary Outcome: Pharmacokinetic Parameter AUC0-∞ of AR-C124910XX
Time Frame: 0, 1, 2, 4, 6, 12, 24, 36, 48 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A | Treatment B | Treatment H
Number analyzed (Participants) | 12 | 13 | 13
ng*h/mL | 1127.8 (39.3) | 1144.2 (36.2) | 1000.4 (33.2)
Statistical Analysis 1: Comparison: Treatment A vs Treatment H; Test type: Other; Ratio of Geometric Least Square Means = 112.73, 90% CI 2-sided [88.61 to 143.42] — Treatment H is the reference treatment
Statistical Analysis 2: Comparison: Treatment B vs Treatment H; Test type: Other; Ratio of Geometric Least Square Means = 114.37, 90% CI 2-sided [91.19 to 143.45] — Treatment H is the reference treatment
Statistical Analysis 3: Comparison: Treatment A vs Treatment B; Test type: Other; Ratio of Geometric Least Square Means = 93.13, 90% CI 2-sided [80.31 to 108.00] — [estimate comment as in outcome 1, analysis 3]

5. Secondary Outcome: Pharmacokinetic Parameter t1/2 of Ticagrelor
Time Frame: 3 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment H
Number analyzed (Participants) | 12 | 13 | 13
hour | 8.303 (1.250) | 8.691 (2.298) | 8.412 (1.248)
Statistical Analysis 1: Comparison: Treatment A vs Treatment H; Test type: Superiority or Other; Mean Difference (Net) = -0.11, 90% CI 2-sided [-0.97 to 0.75] — Treatment A - Treatment H
Statistical Analysis 2: Comparison: Treatment B vs Treatment H; Test type: Superiority or Other; Mean Difference (Net) = 0.28, 90% CI 2-sided [-0.96 to 1.52] — Treatment B - Treatment H
Statistical Analysis 3: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Difference of Least Square Means = -0.36, 90% CI 2-sided [-1.73 to 1.02] — A linear mixed model with sequence, period, and treatment as fixed effects, and subject-within-sequence as a random effect, was used to analyze the natural log-transformed values of the PK parameters. Treatment A - Treatment B

6. Secondary Outcome: Pharmacokinetic Parameter t1/2 of AR-C124910XX
Time Frame: 3 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Treatment A | Treatment B | Treatment H
Number analyzed (Participants) | 12 | 13 | 13
hour | 7.574 (2.079) | 7.596 (1.757) | 8.644 (2.414)
Statistical Analysis 1: Comparison: Treatment A vs Treatment H; Test type: Superiority or Other; Mean Difference (Net) = -1.07, 90% CI 2-sided [-2.62 to 0.48] — Treatment A - Treatment H
Statistical Analysis 2: Comparison: Treatment B vs Treatment H; Test type: Superiority or Other; Mean Difference (Net) = -1.05, 90% CI 2-sided [-2.46 to 0.37] — Treatment B - Treatment H
Statistical Analysis 3: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Difference of Least Square Means = -0.50, 90% CI 2-sided [-1.27 to 0.27] — [estimate comment as in outcome 5, analysis 3]

ADVERSE EVENTS:
Time Frame: Starting from the date of first dose of study medication to follow-up (5-10 days post discharge unit). For HD Subjects, events that occurred during the washout or follow-up periods are attributed to the previous treatment taken.
Arm/Group | Treatment A | Treatment B | Treatment H
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/13 | 0/13
Other Adverse Events (participants affected / at risk) | 2/12 | 3/13 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=12) | Treatment B (N=13) | Treatment H (N=13)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=12) | Treatment B (N=13) | Treatment H (N=13)
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenderness (General disorders) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs shall be entitled to publish or make presentations related to the Study within 2 years of completion of the Study with Sponsor's prior written consent. PIs shall provide the Sponsor with copies of any materials at least thirty (30) days in advance of publication, submission or presentation.

All such publications or presentations shall be consistent with applicable standards, guidelines and laws, not be false or misleading, and not be made for any commercial purpose.